CLINICAL TRIAL: NCT01708122
Title: A Prospective, Randomized, Double Blind Study Comparing the Efficacy and Safety of Fentanyl Nasal Spray to Placebo as an Analgesic, in Patients Undergoing Outpatient Cystoscopic Procedures
Brief Title: Intranasal Fentanyl as an Analgesic for Cystoscopic Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Richard C Reznichek, MD, Medical Doctor, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 13623-01; UL1TR000124 (NIH)
Record Dates: First submitted 2012-03-30; First posted 2012-10-16 (Estimated); Results first posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-07

CONDITIONS: Pain
Keywords: Intranasal fentanyl; Cystoscopy
MeSH Terms: conditions — Pain | interventions — Fentanyl; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fentanyl (Experimental): Subjects will receive either 0.5mL or 1 mL of intranasal fentanyl (50mcg or 100mcg)
  Interventions: Drug: Fentanyl
- Placebo (Placebo Comparator): Subjects will receive either 0.5mL or 1 mL of intranasal saline as placebo.
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Fentanyl — 100 mcg in 1 mL intranasal spray
  Other Names: fentanyl citrate
  Arms: Fentanyl
Drug: saline — Sodium Chloride 0.9% intranasal spray
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of intranasally-administrated fentanyl spray to decrease the pain during cystoscopy (the passage of a telescopic instrument into the bladder for purpose of diagnosing the cause of blood in the urine, urinary complaints or any other problems with the urinary bladder). The current standard practice is to use Lidocaine jelly (a local anesthetic) given through the urethra to lubricate and decrease pain. In this study, an additional medicine (fentanyl) is used to reduce pain that occurs during and after the above procedure.

DETAILED DESCRIPTION:
In this double-blind study, a nasal spray of either the drug (fentanyl -- an opioid analgesic) or placebo (normal saline) is administered before the procedure. There is a 50% chance that patients receive the drug or the placebo. In either case, local Lidocaine jelly is used as an anesthetic in the urethra. Each patient is compensated for time and traveling after the completion of his/her participation.

Patients are asked to arrive between 7 and 11 PM on the evening prior to their procedure for an overnight admission to 5 East ward, on the 5th floor of the Harbor UCLA Medical Center in Torrance, California, United States. Once there, vital signs (blood pressure, pulse, oxygen saturation -- amount of oxygen in the blood, and breathing rate) is checked and an intravenous line is placed. Before, during and after the procedure, patients are asked to rate their pain on a scale of 0 to 10 with 0 being "no pain" and 10 being "the worst pain possible."

Regardless of whether patients are assigned to receive fentanyl or placebo, they receive the standard of care for this cystoscopic procedure.

Once in the cystoscopy room, patients receive the study drug by nasal (into the nose) spray. The study drug is supplied in a pre-filled syringe that contains either 100 mcg of fentanyl or placebo (normal saline with no active medicine in it). Once the study drug is given, the vital signs are closely monitored(checked) until the effect of drug wears off, usually between 2 and 4 hours.

Blood samples are drawn on several occasions. This blood is used to see how much of the study drug (fentanyl or placebo) appears in the blood.

Adverse effects: The well-known adverse effects of opioids may occur after nasal as well as conventional routes of administration; however, severe adverse effects such as respiratory depression or hypotension do not seem to occur in any appreciable frequency.

Intranasal fentanyl has been used safely and effectively in many studies. There are no reports of any serious side effects with the small dose (100 mcg) that is being used in this study. Intranasal fentanyl is generally well tolerated with no serious adverse events. In cancer patients treated for breakthrough pain, the main treatment related side effects were nausea, vertigo, dizziness, constipation, and somnolence. For local side effects, fentanyl displays little local irritation, nasal discomfort or taste experiences. Nasal irritation, skin pain, nasal mucosa ulcers and dysgeusia have been occasionally reported as minor side effects.

The following minor side effects have been reported with other forms of fentanyl (oral, patch or intravenous): anxiety; confusion; difficulty walking; dizziness; drowsiness; dry mouth; headache; itching; nausea and vomiting.

The following severe side effects have not been reported with intranasal fentanyl but have been reported with other forms of fentanyl (oral, patch or intravenous): allergic reactions (rash; hives; difficulty breathing; tightness in the chest; swelling of the mouth, face, lips, or tongue); excessive dizziness; excessive drowsiness; fainting; fatigue; hallucinations; muscle rigidity; seizures; shock (changes in skin color); slow heartbeat; respiratory depression or slowed breathing; trouble breathing and feeling of weakness.

Advantages to patients: If effective, less pain during and after the cystoscopic procedure and better tolerance of the procedure.

Advantages to humanity: If effective, nasal fentanyl could be used as a means to reduce pain before and during cystoscopic procedures.

These benefits may not happen and unexpected side effects may develop.

ELIGIBILITY:
Inclusion Criteria:

1. Urological indications for cystoscopic procedure.

Exclusion Criteria:

1. History of analgesia abuse or former opioid addiction.
2. Allergy to fentanyl.
3. Acute/chronic nasal problems such as rhinitis or sinusitis.
4. Positive urine pregnancy test / lactation.
5. Acute bronchial asthma / upper airway obstruction.
6. Presence of bradycardia or a history of seizures.
7. Concomitant use of drugs that inhibit CYP3A4 (e.g., ritonavir, ketoconazole, itraconazole, troleandomycin, clarithromycin, nelfinavir, nefazodone, amprenavir, aprepitant, diltiazem, erythromycin, fluconazole, fosamprenavir, MAO inhibitors and verapamil)
8. 0-10 NRS pain score more than 3 on baseline.
9. Any situation or condition which, in the investigator's opinion, puts the subject at significant risk, or could confound the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2009-05; Primary Completion 2013-03 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Reznichek, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Harbor UCLA Medical Center Urology Clinic, Torrance, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seventy-one patients agreed to participate in the study and signed informed consent. Nine patients declined to proceed. Seven did not pass pre-anesthesia screening due to pre-existing medical conditions. Cystoscopic procedures were deemed no longer indicated for two patients. Ultimately, 53 patients were randomized and completed the study.
Groups:
- Placebo: Subjects will receive 0.1 mL of intranasal saline as placebo.
  saline: Sodium Chloride 0.9% intranasal spray
- Fentanyl: Subjects receiving either 50mcg or 100mcg
Period: Overall Study
Arm/Group | Placebo | Fentanyl
Started | 27 | 26
Completed | 27 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fentanyl: Subjects will receive 50 to 100 mcg intranasal fentanyl
  Fentanyl: 100 mcg in 1 mL intranasal spray
- Placebo: Subjects will receive intranasal saline as placebo.
  Saline: Sodium Chloride 0.9% intranasal spray
- Total: Total of all reporting groups
Arm/Group | Fentanyl | Placebo | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Mean (Full Range); unit: years] | 45.2 [21 to 65] | 47.1 [29 to 74] | 46.2 [21 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 14 | 11 | 25
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Pre Procedure 0 - 10 Pain Numerical Rating Scale
Description: The NRS pain assessment (0 = no pain to 10 = worst possible pain) is recorded as outlined below:
  1. baseline pain score at admission, when the subject checks in, 2 Upon entry of the cystoscope into the urethral meatus, 3. and thirty minutes after the cystoscopic procedure has been completed.
Time Frame: Pre procedure, During procedure, Post procedure
Measure: Median (Full Range); unit: 0 - 10 Pain Numerical Rating Scale
Arm/Group | Fentanyl | Placebo
Number analyzed (Participants) | 26 | 27
0 - 10 Pain Numerical Rating Scale
  Pre-procedure | 0 [0 to 7] | 0 [0 to 6]
  During procedure | 7 [0 to 10] | 5 [0 to 10]
  Post Procedure | 0 [0 to 7] | 0 [0 to 10]

2. Secondary Outcome: O2 Saturation Post Drug Administration
Description: After administration of the study drug, the subject is monitored (oxygen saturation), for any signs of respiratory depression or the presence of complications or side-effects including apnea or oxygen desaturation.
Time Frame: Baseline, 5 minutes 10 minutes and 30 minutes post drug-administration.
Measure: Mean (Full Range); unit: percentage of O2 Saturation
Arm/Group | Fentanyl | Placebo
Number analyzed (Participants) | 26 | 27
percentage of O2 Saturation
  Baseline | 99.4 [96 to 100] | 99.3 [96 to 100]
  5 minutes | 99.3 [97 to 100] | 99.3 [96 to 100]
  10 Minutes | 99.5 [97 to 100] | 99.4 [96 to 100]
  30 Minutes | 99.3 [96 to 100] | 99.4 [96 to 100]

ADVERSE EVENTS:
Time Frame: From administration of study drug until 3 hours post administration
Description: By direct questioning regarding the presence of the following: Nasal Irritation, nausea, vomiting, dizziness, respiratory distress, confusion, headache, dry mouth and any other discomfort no related to the surgical procedure with the possible answers yes or no. Subject can also report spontaneously during their stay in the department.
Groups:
- Fentanyl: Subjects receiving either 0.5mL or 1 mL of intranasal fentanyl (50mcg or 100mcg)
  Fentanyl: 100 mcg in 1 mL intranasal spray
- Placebo: Subjects receiving either 0.5mL or 1 mL intranasal saline as placebo.
  Saline: Sodium Chloride 0.9% intranasal spray
Arm/Group | Fentanyl | Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 9/26 | 4/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fentanyl (N=26) | Placebo (N=27)
Nausea (General disorders) | 2 (2) | 1 (1)
Dizziness (General disorders) | 2 (2) | 0 (0)
headache (General disorders) | 1 (1) | 2 (2)
Nasal Irritation (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No